CLINICAL TRIAL: NCT03030976
Title: An Open-labeled, Uncontrolled, Single-arm Pilot Study to Evaluate Cellular Immunotherapy Using CD19-targeted Chimeric Antigen Receptor Engineered T Cells in Patients With CD19+ B Cell Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of CD19 Redirected Autologous T Cells for CD19 Positive Systemic Lupus Erythematosus (SLE)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai GeneChem Co., Ltd. (Industry)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CART for SLE
Record Dates: First submitted 2017-01-22; First posted 2017-01-25 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: CD19; CAR-T; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduce B cells (Experimental): Patients receive cyclophosphamide to reduce B cells before CD19-CART infusion. It will also reduce the side effects of cell damage due to antitumor activity.
  Interventions: Drug: cyclophosphamide
- Treatment of SLE (Experimental): Patients receive anti-CD19-CAR-T cells to treatment of SLE. The purpose of this study is to assess the safety and efficacy of CD19 CAR-T cells in the treatment of SLE.
  Interventions: Drug: anti-CD19-CAR-T cells

INTERVENTIONS:
Drug: cyclophosphamide — Patients receive cyclophosphamide (Cy) on day -2 and day -1 to reduce B cells. The dose is 0.5g/m2/d.
  Other Names: Cy
  Arms: Reduce B cells
Drug: anti-CD19-CAR-T cells — A 2nd CAR, CD19 as target protein, 4-1BB as co-stimulator, and optimized the spatial conformation by a suitable hinge & transmembrane domain sequences. Patients infused with anti-CD19-CAR-T cells transduced with lentivirus on day 0 in the absence of disease progression or unacceptable toxicity to treatment of SLE. The dose is 1E6~1E7 CD19-CAR positive T cells. The cells infusion process may last for 30 min.
  Other Names: 2nd CAR-T
  Arms: Treatment of SLE

SUMMARY:
CAR-T therapy was therefore proposed and has been recently used for cancer treatment. It has been hailed for its promising remission rates after early stage clinical trials for acute lymphoblastic leukemia. However, CAR-T therapy is seldom used for autoimmune diseases. Researchers only use it for the treatment of multiple sclerosis (MS, an autoimmune disease of the central nervous system). SLE is a kind of autoimmune diseases which involving multiple systems, organs and with the present of a variety of autoantibodies. In the conventional treatment options, SLE could be treated with chemotherapy drugs or hormone drugs. But chemotherapy and hormone drugs could barely cured SLE. And now, chimeric antigen receptor modified T cell infusion maybe an effective treatment to solve these problems. The investigators use a 2nd CAR- T with the optimized hinge and transmembrane domain to treat patients with SLE. The purpose of this study is to assess the safety and efficacy of this 2nd CAR-T cells in the treatment of SLE.

DETAILED DESCRIPTION:
This study is being conducted to assess anti-CD19-CAR-T cells safety and efficacy in treating patients with systemic lupus erythematosus（SLE）.The investigators constructed a 2nd CAR, using CD19 as target, using 4-1BB as co-stimulator, and optimized the spatial conformation by a suitable hinge and transmembrane domain sequences. The infusion dose is (1-10)E6 CAR positive T cells/kg, and the specific cells numbers depends on the situation of individual CAR-T cells preparation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of systemic lupus erythematosus (SLE) patients
* Patients with CD19+ B-cell SLE as confirmed by Flow Cytometry
* Age: 18-69 years old
* Creatinine < 1.5 mg/dl
* cardiac ejection fraction>55%
* hemoglobin>9g/dL
* Bilirubin <2.0 mg/dl
* Successful test expansion of T-cells
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled active infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates<5% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, serious arrhythmia)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Safety of CAR-T cell（i.v.）by number of patients with adverse event | 6 weeks
  adverse event is evaluated with CTCAE, version 4.0

SECONDARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  summarize tumor response by overall response rates
3. Detection of transferred T cells in the circulation using quantitative -PCR | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Guo, Doctor, Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided